CLINICAL TRIAL: NCT03307239
Title: Efficacy of Cold Application on Pain During Chest Tube Removal: A Randomized Controlled Trial : A CONSORT Compliant Article
Brief Title: Cold Application on Pain During Chest Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103044
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Chest Tube Removal

STUDY DESIGN:
Intervention Model Description: subjects in the experimental group received cold application of 600 g ice packs 15 min before CTR, whereas subjects in the sham group
Who Masked: Participant
Masking Description: the researcher assigned participants to one of the two groups: cold application (experimental group) or tap water packs application (sham group) according the random allocation sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold application (experimental group) (Experimental): subjects in the experimental group (n = 30) received cold application of 600 g ice packs 15 minutes before CTR
  Interventions: Other: cold application
- tap water packs application (sham group) (Sham Comparator): subjects in the sham group (n = 30) received tap water packs.
  Interventions: Other: tap water packs application

INTERVENTIONS:
Other: cold application — We manufactured two ice packs (17 × 12 cm) with a combined weight of 600 g. The ice packs were inserted into adjustable wraps made in our hospital so that they can be fixed next to the skin on each side of the chest tube in patients awaiting CTR. The combined contact area of the ice packs was approximately 25 cm in diameter around the chest tube.
  For patients of the experimental group, they were received 15-minutes cold application.
  Arms: cold application (experimental group)
Other: tap water packs application — We manufactured two tap water packs (17 × 12 cm) with a combined weight of 600 g. The tap water packs were inserted into adjustable wraps made in our hospital so that they can be fixed next to the skin on each side of the chest tube in patients awaiting CTR. The combined contact area of the tap water packs was approximately 25 cm in diameter around the chest tube.
  For patients of the sham group, they were received 15-minutes tap water application.
  Arms: tap water packs application (sham group)

SUMMARY:
Abstract Objectives: Use of analgesics is the most common method to alleviate the pain induced by chest tube removal (CTR), but patient response to medication can vary and may not be achieved complete relaxation. This study was to determine the effectiveness of cold application in combination with standard analgesic administration before CTR on CTR-induced pain.

Methods: A prospective, randomized, single-blind, placebo sham-controlled study was conducted. In addition to the same routine care, subjects in the experimental group (n = 30) received cold application of 600 g ice packs 15 minutes before CTR, whereas subjects in the placebo sham group (n = 30) received tap water packs. Numerical rating scale was used to measured pain intensity before, immediately after, and 10 minutes after CTR.

ELIGIBILITY:
Inclusion Criteria:

* (a) age greater than 20 years, (b) single chest-tube insertion, (c) first-time insertion of the chest tube, (d) ability to verbally report pain, (e) body mass index of < 30 kg/m2, and (f) normal vital signs.

Exclusion Criteria:

* cold urticaria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS) | before cold application
  the intensity of pain at the chest tube replacement
numerical rating scale (NRS) | immediately after chest tube removal
  the intensity of pain at the chest tube removal
numerical rating scale (NRS) | 10 minutes after chest tube removal
  the intensity of pain at the chest tube removal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh LY, Chen YR, Lu MC. Efficacy of cold application on pain during chest tube removal: a randomized controlled trial: A CONSORT-compliant article. Medicine (Baltimore). 2017 Nov;96(46):e8642. doi: 10.1097/MD.0000000000008642. PMID 29145288